CLINICAL TRIAL: NCT02073812
Title: A Phase 1, Randomized, Open-Label, Trial Evaluating the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations of Intravenous Carbavance™ (RPX2014/RPX7009) in Healthy Adult Subjects
Brief Title: Evaluating the Plasma, Epithelial Lining, and Alveolar Macrophage Concentrations of Intravenous Carbavance™ (RPX2014/RPX7009) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rempex 503
Record Dates: First submitted 2014-02-14; First posted 2014-02-27 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — RPX7009

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple dose of Carbavance (RPX7009/RPX2014) (Experimental): Multiple dose of Carbavance
  Interventions: Drug: RPX7009 and RPX2014

INTERVENTIONS:
Drug: RPX7009 and RPX2014 — The study is designed to enroll approximately 25 healthy subjects. The study will evaluate the plasma, epithelial lining fluid, and alveolar macrophage concentrations of Carbavance (RPX7009/RPX2014)

SUMMARY:
RPX7009(beta-lactamase inhibitor) is being studied in combination with a carbapenem (RPX2014) to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem (RPX2014) plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the pharmacokinetics of intravenous RPX2014 and RPX7009 in plasma and epithelial fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females, 18 to 55 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 30 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive) at the time of screening.
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms (ECGs), physical examination) as deemed by the PI.
4. Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to Day 1.
5. Voluntarily consent to participate in the study.

Exclusion Criteria:

1. History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug/alcohol testing at screening (or Day -1).
3. Positive testing for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg).
4. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
5. Hypersensitivity or idiosyncratic reaction to beta-lactam antibiotics (e.g. penicillins, cephalosporins, carbapenems, etc.).
6. Clinically significant pulmonary or any other disease that prevents a subject from undergoing bronchoscopy with bronchopulmonary lavage.
7. History of seizures (e.g., epilepsy), head injury or meningitis requiring ongoing anti-seizure medications.
8. Use of any prescription medication (with the exception of hormonal contraceptives or hormone replacement therapy for females) within 14 days prior to Day 1.
9. Participation in another investigational clinical trial within 30 days prior to Day 1.
10. Females who are pregnant or lactating.
11. Surgery within the past three months prior to Day 1 determined by the PI to be clinically relevant.
12. Any acute illness including clinically significant infection within 30 days prior to Day 1.
13. QTcF interval >450 msec, or history of prolonged QT syndrome at screening (or Day 1).
14. Calculated creatinine clearance less than 80 mL/min (Cockroft-Gault method) at screening.
15. Subjects who have any clinically significant abnormalities on laboratory values at screening (or Day -1), including:

    1. White blood cell count (WBC) < 3,000/mm3, hemoglobin < 11g/dL.
    2. Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
16. Liver function abnormalities at screening (or Day -1) (defined by an elevation in bilirubin, AST or ALT 1.5 x ULN of the normal range for subjects based on age and sex).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics from baseline through the end of the study | 2 days
  Assessment of plasma, ELF and AM concentrations of RPX2014 and RPX7009 after 3 doses of Carbavance

SECONDARY OUTCOMES:
IV Carbavance concentrations in lung fluid | 2 days
  Plasma, ELF and AM concentrations of intravenous Carbavance in healthy adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gotfried, MD, Principal Investigator — Pulmonary Associates
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States